CLINICAL TRIAL: NCT05024006
Title: An International Randomized Trial of Additional Treatments for COVID-19 in Hospitalized Patients Who Are All Receiving the Local Standard of Care Philippines
Brief Title: Public Health Emergency: SOLIDARITY TRIAL Philippines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Philippines (Other)
Responsible Party: Principal Investigator, Marissa Alejandria MD, Professor, University of the Philippines
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SJREB-2020-20
Record Dates: First submitted 2021-08-21; First posted 2021-08-27 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Covid19
Keywords: Solidarity; Hydroxychloroquine; Lopinavir+Ritonavir; Interferon Beta 1a; Remdesivir
MeSH Terms: conditions — COVID-19 | interventions — remdesivir; Hydroxychloroquine; Lopinavir; Interferon beta-1a; acalabrutinib

STUDY DESIGN:
Intervention Model Description: Adaptive design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- LSoC (No Intervention): Local Standard of Care
- Rem+LSoC (Experimental): Remdesivir with Local Standard of Care
  Interventions: Drug: Remdesivir
- HCQ+LSoC (Experimental): Hydroxychloroquine with Local Standard of Care
  Interventions: Drug: Hydroxychloroquine
- Lopi/Rito+LSoC (Experimental): Lopinavir/Ritonavir with Local Standard of Care
  Interventions: Drug: Lopinavir / Ritonavir
- Lopi/Rito+IFN+LSoC (Experimental): Lopinavir/Ritonavir and Interferon Beta 1a with Local Standard of Care
  Interventions: Drug: Lopinavir / Ritonavir; Drug: Interferon beta-1a
- IFN+LSoC (Experimental): Interferon Beta 1a with Local Standard of Care
  Interventions: Drug: Interferon beta-1a
- ACB+LSoC (Experimental): Acalabrutinib with Local Standard of Care
  Interventions: Drug: Acalabrutinib

INTERVENTIONS:
Drug: Remdesivir — Two intravenous loading doses, then daily infusion for 10 days
  Arms: Rem+LSoC
Drug: Hydroxychloroquine — Two oral loading doses, then orally twice daily for 10 days
  Arms: HCQ+LSoC
Drug: Lopinavir / Ritonavir — Orally twice daily for 14 days
  Arms: Lopi/Rito+IFN+LSoC; Lopi/Rito+LSoC
Drug: Interferon beta-1a — Daily injection for 6 days
  Arms: IFN+LSoC; Lopi/Rito+IFN+LSoC
Drug: Acalabrutinib — Orally twice daily for 10 days
  Arms: ACB+LSoC

SUMMARY:
This study is an adaptive, randomized, open-label, controlled clinical trial utilizing an adaptive design to compare effects of repurposed drugs with local standard of care alone on major inpatient hospital outcomes. This is performed worldwide in collaboration with WHO.

ELIGIBILITY:
Inclusion Criteria:

* Consenting adults (age ≥18) hospitalised with the following criteria will be included in the study:

  1. Probable or confirmed COVID-19 regardless of severity, i.e., mild, moderate and severe cases
  2. Not already receiving any of the study drugs
  3. Without known allergy or contraindications to any of the study drugs (in the view of the physician responsible for their care), and
  4. Without anticipated transfer within 72 hours to a non-study hospital.

Exclusion Criteria:

* Patients with contraindications to any of the study drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1314 (Actual)
Dates: Start 2020-04-23 (Actual); Primary Completion 2021-04-17 (Actual); Study Completion 2021-04-17 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | Number of days from hospital admission up to 28 days post discharge

SECONDARY OUTCOMES:
Duration of hospital stay | Number of days from hospital admission to discharge up to 28 days post admission
Time to first receiving ventilation | Number of days from hospital admission to day of receiving ventilatory support up to 28 days post admission

CONTACTS AND LOCATIONS:
Locations (25):
- Philippines (25):
  - Baguio General Hospital, Baguio City, Benguet
  - Cebu Doctor's University Hospital, Cebu City, Cebu
  - Perpetual Succor Hospital Cebu, Cebu City, Cebu
  - Vicente Sotto Memorial Medical Center, Cebu City, Cebu
  - Southern Philippines Medical Center, Davao City, Davao Region
  - West Visayas University Medical Center, Iloilo City, Iloilo
  - St Luke's Medical Center Global, City of Taguig, National Capital Region
  - Makati Medical Center, Makati City, National Capital Region
  - Chinese General Hospital, Manila, National Capital Region
  - Manila Doctors Hospital, Manila, National Capital Region
  - ManilaMed - Medical Center Philippines, Manila, National Capital Region
  - San Lazaro Hospital, Manila, National Capital Region
  - UP - Philippine General Hospital, Manila, National Capital Region
  - Asian Hospital and Medical Center, Muntinlupa, National Capital Region
  - Research Institute for Tropical Medicine, Muntinlupa, National Capital Region
  - San Juan de Dios Educational Foundation Inc - Hospital, Pasay, National Capital Region
  - The Medical City, Pasig, National Capital Region
  - Diliman Doctors Hospital, Quezon City, National Capital Region
  - Fe Del Mundo Medical Center, Quezon City, National Capital Region
  - Lung Center of the Philippines, Quezon City, National Capital Region
  - St Luke's Medical Center Quezon City, Quezon City, National Capital Region
  - University of the East Ramon Magsaysay Memorial Medical Center, Quezon City, National Capital Region
  - World Citi Medical Center, Quezon City, National Capital Region
  - Cardinal Santos Medical Center, San Juan City, National Capital Region
  - Batangas Medical Center, Batangas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grundeis F, Ansems K, Dahms K, Thieme V, Metzendorf MI, Skoetz N, Benstoem C, Mikolajewska A, Griesel M, Fichtner F, Stegemann M. Remdesivir for the treatment of COVID-19. Cochrane Database Syst Rev. 2023 Jan 25;1(1):CD014962. doi: 10.1002/14651858.CD014962.pub2. PMID 36695483